CLINICAL TRIAL: NCT06635577
Title: Changing Quantitative Reasoning Across Development
Brief Title: Modifying Cognitive Strategies for Comparing Proportions
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Hurst, PhD (Other)
Collaborators: Rutgers, The State University of New Jersey (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Michelle Hurst, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2023001794; R00HD104990 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Proportional Reasoning
Keywords: proportions; mathematical concepts; strategy use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proportion Judgements (Experimental): This is the sole arm of the study. All participants will be observed under normal conditions and then those same participants will undergo a behavioral intervention.
  Interventions: Behavioral: Verbal Interference Task

INTERVENTIONS:
Behavioral: Verbal Interference Task — During the second half of the study, participants will undergo an interference task such as repetition of the word "the"; or shadowing a radio broadcast in order to increase cognitive load and disrupt the use of a mental workspace.

SUMMARY:
The goal of this study is to understand the cognitive processes underlying quantitative and relational reasoning, including the understanding of mathematical information (e.g., numbers, proportions, percentages, geometry) and related relational concepts (e.g., analogies, the concepts same/different), as well as how people's reasoning can be changed by external factors. The main question it aims to answer is:

How does the introduction of a secondary task affect the behavior of children and adults when reasoning about proportions in different formats? Participants will be asked to make judgements about images with and without the presence of a distractor task.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing people within the target age range (either 8-years-old OR 18- to 64-years-old) for the study version

Exclusion Criteria:

* Individuals with known developmental or cognitive disorders
* Participants or parents of participants must speak/read sufficient English to read and complete the informed consent document

Ages: 7 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Overall Performance | After enrollment in a single study session
  A proportion correct will be calculated, with a score closer to 1 indicating more questions answered correctly. Reaction time will also be tracked, with a faster reaction time indicating ease and/or efficiency with the task.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Center for Cognitive Science, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participant responses to all measures, as well as de-identified demographics (e.g., age, gender) will be made publicly available on a data repository.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning when the results are published (if not earlier) with no planned end date
Access Criteria: De-identified data will be publicly available under a creative commons license only requesting attribution.

REFERENCES:
- [Background] Boyer TW, Levine SC, Huttenlocher J. Development of proportional reasoning: where young children go wrong. Dev Psychol. 2008 Sep;44(5):1478-90. doi: 10.1037/a0013110. PMID 18793078
- [Background] Hurst MA, Piantadosi ST. Continuous and discrete proportion elicit different cognitive strategies. Cognition. 2024 Nov;252:105918. doi: 10.1016/j.cognition.2024.105918. Epub 2024 Aug 16. PMID 39153444

DOCUMENTS (1):
  • Informed Consent Form (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT06635577/ICF_000.pdf